CLINICAL TRIAL: NCT05325450
Title: Optimization of Hearing Performance in the Subject Implanted With Profound Asymmetric Deafness
Brief Title: Optimization of Hearing Performance in the Subject Implanted
Acronym: OPERSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RC31/21/0125
Record Dates: First submitted 2022-03-01; First posted 2022-04-13 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Hearing Loss
Keywords: deafness, cochlear implant
MeSH Terms: conditions — Hearing Loss; Deafness | interventions — Medicare Part A

STUDY DESIGN:
Intervention Model Description: two within-subject crossover experiments (short-term and long-term) where each subject will follow two phases of the protocol (training A and training B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training A (Experimental): Training A in Unilaterally postlingually-deafened adult cochlear implanted candidates
  Interventions: Procedure: Program A
- Training B (Experimental): Training B in Unilaterally postlingually-deafened adult cochlear implanted candidates
  Interventions: Procedure: Program B
- Control (Active Comparator): Training in bilaterally postlingually-deafened adult cochlear implanted candidates
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Program A — Presentation of the sentence to the implant alone
  Arms: Training A
Procedure: Program B — Presentation of the sentence to the implanted ear, associated for the non-implanted ear
  Arms: Training B
Procedure: Control — Presentation of the sentences alternately to the most recently implanted ear and both implanted ears at the same time
  Arms: Control

SUMMARY:
In the past two decades, the selection criteria for cochlear implantation have been greatly relaxed so that about 60-70% of present cochlear implant (CI) candidates have significant residual hearing in their contralateral ear. However, contralateral hearing is often not considered in rehabilitation programs, mainly due to the lack of scientific evidence on the role it may play. The present project aims to better understand the mechanisms of perceptual learning of CI-processed speech after implantation and to develop and test rehabilitation strategies for CI users.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Unilaterally postlingually-deafened adult cochlear implanted candidates (IC-Uni)
* Person with almost normal or moderate contralateral hearing ( under 60dB)
* Cochlear implanted person whose activation has not yet been performed
* Cochlear implanted subjects with bilateral post-lingual profound deafness, who already benefit from a unilateral cochlear implant and candidates to a bilateral cochlear implant
* Affiliated to social security

Exclusion Criteria:

* - Subjects under juridical protections or tutelage measure
* Subjects with associated neurological or neurodegenerative conditions
* Significant anatomical changes on CT scan of the temporal bone that may interfere with the insertion of the cochlear implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-01-18 (Estimated); Study Completion 2025-01-18 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the percentage of correct speech recognition after training between the two training programs | Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Marx, Toulouse, France

IPD SHARING:
Plan to Share IPD: No